CLINICAL TRIAL: NCT02253303
Title: Evaluation of the Extraction-site Location in Laparoscopic Colorectal Surgery - Midline Incision vs Off-midline Incision-
Brief Title: Evaluation of the Extraction-site, - Midline Incision vs Off-midline Incision-
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hiroki Yamaue (Other)
Collaborators: Katsunari Takifuji (Unknown)
Responsible Party: Sponsor-Investigator, Hiroki Yamaue, Chief and professor of second department of surgery, Wakayama Medical University
Organization: Wakayama Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WMU1398
Record Dates: First submitted 2014-09-24; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Midline incision (Experimental): The extraction-site incision in laparoscopic colectomy is middline
  Interventions: Other: midline incision or off-midline incision
- off-midline incision (Active Comparator): The extraction-site incision in laparoscopic colectomy is off-middline
  Interventions: Other: midline incision or off-midline incision

INTERVENTIONS:
Other: midline incision or off-midline incision — Eligible patients are randomized to midline incision or off-midline incision group in laparoscopic colectomy

SUMMARY:
The purpose of this study is to evaluate the midline extraction incision in patients with colon cancer. A prospective randomized controlled trial is conducted to compare midline extraction incision with off-midline extraction incision.

DETAILED DESCRIPTION:
Laparoscopic colon surgery is less invasive and more cosmetic than open surgery. But the extraction-site incision is 4 to 5 cm, and it is the largest and most painful incision in laparoscopic colon surgery. The purpose of this study is to evaluate the midline extraction incision in patients with colon cancer. A prospective randomized controlled trial is conducted to compare midline extraction incision with off-midline extraction incision. The investigators hypothesize that the use of the midline extraction incision in laparoscopic colon surgery will result in more cosmetic effect and better quality of life compared to the off-midline extraction incision.

ELIGIBILITY:
Inclusion Criteria:

* Tumor size is less than 5cm
* No history of laparotomy
* No bowel obstruction by tumor

Exclusion Criteria:

* Patients who can't respond to medical question
* Patients who receive steroids or insulin therapy
* Uncontrolled DM
* Severe respiratory failure(HOT)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
cosmetic effect | 1 year
  Scar assessment score on the patient and observer scar assessment scale(POSAS)

SECONDARY OUTCOMES:
Quality of life | 7 days, 14 days and 30 days
  Questionnaire on the SF-36 v2 acute

OTHER OUTCOMES:
Incisional hernia | 1 year
  Numbers of participants with incisional hernia

CONTACTS AND LOCATIONS:
Overall Officials: HIroki Yamaue, Chief prof., Study Director — Second Department of Surgery, Wakayama Medical University

REFERENCES:
- [Background] Samia H, Lawrence J, Nobel T, Stein S, Champagne BJ, Delaney CP. Extraction site location and incisional hernias after laparoscopic colorectal surgery: should we be avoiding the midline? Am J Surg. 2013 Mar;205(3):264-7; discussion 268. doi: 10.1016/j.amjsurg.2013.01.006. Epub 2013 Jan 31. PMID 23375702
- [Background] Singh R, Omiccioli A, Hegge S, McKinley C. Does the extraction-site location in laparoscopic colorectal surgery have an impact on incisional hernia rates? Surg Endosc. 2008 Dec;22(12):2596-600. doi: 10.1007/s00464-008-9845-8. Epub 2008 Mar 18. PMID 18347858
- [Background] Lee L, Mappin-Kasirer B, Sender Liberman A, Stein B, Charlebois P, Vassiliou M, Fried GM, Feldman LS. High incidence of symptomatic incisional hernia after midline extraction in laparoscopic colon resection. Surg Endosc. 2012 Nov;26(11):3180-5. doi: 10.1007/s00464-012-2311-7. Epub 2012 May 12. PMID 22580878